CLINICAL TRIAL: NCT02922582
Title: A Randomized, Single-Blind, Active-Controlled, Dose-Ranging Study to Evaluate the Pharmacokinetics, Safety, and Efficacy of Local Administration of DepoTXA for Reduced Postsurgical Bleeding in Subjects Undergoing Total Knee Arthroplasty
Brief Title: Study of Local Administration of DepoTXA for Reduced Postsurgical Bleeding in Subjects Undergoing TKA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 404-C-201
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- DepoTXA 400mg (Experimental): 400mg Intracapsular at the end of surgery one time
  Interventions: Drug: DepoTXA
- DepoTXA 800mg (Experimental): 800mg Intracapsular at the end of surgery one time
  Interventions: Drug: DepoTXA
- DepoTXA 1200mg (Experimental): 1200mg Intracapsular at the end of surgery one time
  Interventions: Drug: DepoTXA
- IV Tranexamic acid (TXA) (Active Comparator): 1 g of IV TXA at the end of surgery
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: DepoTXA
  Arms: DepoTXA 1200mg; DepoTXA 400mg; DepoTXA 800mg
Drug: Tranexamic Acid
  Arms: IV Tranexamic acid (TXA)

SUMMARY:
This is a Phase 2, randomized, single-blind, active-controlled dose-ranging study in subjects scheduled to undergo total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Approximately 60 subjects (15 per arm) are planned for enrollment. Subjects will be randomized in a 1:1:1:1 ratio to receive either DepoTXA 400 mg, DepoTXA 800 mg, DepoTXA 1200 mg, or IV TXA (Cyklokapron® 1 gram).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years of age at screening.
2. Scheduled to undergo elective unilateral open TKA under general, spinal, or regional anesthesia.
3. American Society of Anesthesiology (ASA) physical status 1, 2, or 3.
4. Female subject must be surgically sterile; or at least 2 years postmenopausal; or have a monogamous partner who is surgically sterile; or practicing double-barrier contraception; or practicing abstinence (must agree to use double-barrier contraception in the event of sexual activity); or using an insertable, injectable, or transdermal, contraceptive approved by the FDA for greater than 2 months prior to screening and commit to the use of an acceptable form of birth control for the duration of the study and for 30 days after completion of the study.
5. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration.
2. Planned concurrent surgical procedure (e.g., bilateral TKA).
3. Prior open knee surgery on ipsilateral knee. Prior arthroscopy is permitted.
4. Subjects taking a medication with a known procoagulant effect (e.g., combination hormonal contraceptives, Factor IX complex concentrates or anti-inhibitor coagulant concentrates, or all-trans retinoic acid).
5. Contraindication or hypersensitivity to TXA.
6. History of thrombosis or prior Venous thromboembolism (VTE).
7. Known coagulopathy or active intravascular clotting.
8. Prior myocardial infarction.
9. Prior cardiovascular accident (stroke) or subarachnoid hemorrhage.
10. History of epilepsy.
11. Presence of an intravascular stent.
12. History of impaired kidney function, chronic respiratory disease, rheumatoid arthritis, coagulopathy, or loss of sensation in extremities.
13. Renal insufficiency (serum creatinine level >2 mg/dL).
14. Anemia (Hb level <10 g/dL).
15. Uncontrolled anxiety, psychiatric, or neurological disorder that might interfere with study assessments.
16. Acquired defective color vision.
17. Malignancy in the last 2 years, with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
18. Suspected or known history of drug or alcohol abuse within the previous year.
19. Body weight <50 kg (110 pounds) or a body mass index >44 kg/m2.
20. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Danesi, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (5):
- United States (5):
  - Ortho Arizona, Gilbert, Arizona
  - University of Miami Hospital, Miami, Florida
  - Kendall Regional Medical Center, Miami, Florida
  - Ohio State University/Wexner Medical Center, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between October 28, 2016 and October 12, 2017 at 4 US sites. The study was terminated on 27-Nov-2017 due to low enrollment.
Pre-assignment Details: One patient was screened but was not randomized due to not meeting inclusion criteria.
Groups:
- DepoTXA 400mg: Single injection of DepoTXA 400 mg into the joint space via catheter prior to capsular closure
- DepoTXA 800mg: Single injection of DepoTXA 800 mg into the joint space via catheter prior to capsular closure
- DepoTXA 1200mg: Single injection of DepoTXA 1200 mg into the joint space via catheter prior to capsular closure
Period: Overall Study
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Started | 4 | 4 | 4 | 4
Completed | 4 | 3 | 4 | 4
Not Completed | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: All subjects who received study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA) | Total
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7.12) | 66 (1.73) | 59.3 (5.38) | 58.0 (6.16) | 61.8 (6.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 2 | 9
  Male | 1 | 1 | 2 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 4 | 4 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 3 | 3 | 3 | 3 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-versus-time Curve From Time 0 Extrapolated to Infinity After Drug Administration
Time Frame: Baseline; 5, 15, and 30 min; at 1, 2, 4, 6, 8, 12, 16, and 24 hours after study drug administration for all treatment groups. Additional blood samples were collected at 36, 48, 60, 72, and 96 hours for DepoTXA-treated subjects.
Population: Pharmacokinetic (PK) analysis set: All subjects who received study drug, provided sufficient samples to allow for calculation of PK parameters required for analysis, and who did not have significant protocol deviations
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 2 | 4 | 4
hr*ng/mL | 46462.15 (6935.828) | 106422.7 (42128.84) | 148806.2 (14137.74) | 134602.2 (29975.88)

2. Primary Outcome: Area Under the Plasma Concentration-versus-time Curve From Time 0 to the Last Collection Time After Drug Administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 2 | 4 | 4
hr*ng/mL | 43784.71 (6463.220) | 104546.5 (42813.20) | 143562.9 (13931.94) | 131153.0 (27286.97)

3. Primary Outcome: Maximum Plasma Concentration (Cmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 2 | 4 | 4
ng/mL | 2775.0 (741.96) | 7722.0 (2015.25) | 9827.0 (1545.83) | 125390.0 (154587.6)

4. Primary Outcome: Time to Maximum Plasma Concentration (Tmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 2 | 4 | 4
hr | 1.6 (0.55) | 1.5 (0.57) | 2.5 (0.96) | 0.1 (0)

5. Primary Outcome: The Apparent Terminal Elimination Rate Constant
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 2 | 4 | 4
1/hr | 0.048 (0.0084) | 0.035 (0.0120) | 0.035 (0.0095) | 0.136 (0.0261)

6. Primary Outcome: The Apparent Terminal Elimination Half-life
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 2 | 4 | 4
hr | 14.679 (2.6980) | 21.132 (7.2508) | 20.956 (5.7276) | 5.220 (0.8540)

7. Secondary Outcome: Summary of Neurological Assessments (Proportion of Subjects Who Were Oriented and Proportion of Subjects Who Had Any of the Neurologic Events) at Each Assessed Timepoint
Description: Neurological assessment at 12, 24, 36, 48, 60, 72, and 96 hours after study drug administration
Time Frame: 12, 24, 36, 48, 60, 72, and 96 hours after study drug administration
Population: Safety analysis set: All subjects who received study drug treatment
Measure: Number; unit: participants
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 3 | 4 | 4
participants
  Number of subjects who had any of the neurologic events at baseline | 0 | 0 | 0 | 0
  Number of subjects who had any of the neurologic events at 12 hours | 0 | 0 | 0 | 0
  Number of subjects who had any of the neurologic events at 24 hours | 0 | 0 | 0 | 0
  Number of subjects who had any of the neurologic events at 36 hours | 0 | 0 | 0 | 0
  Number of subjects who had any of the neurologic events at 48 hours | 0 | 0 | 0 | 0
  Number of subjects who had any of the neurologic events at 60 hours | 0 | 0 | 0 | 0
  Number of subjects who had any of the neurologic events at 72 hours | 0 | 0 | 0 | 0
  Number of subjects who had any of the neurologic events at 96 hours | 0 | 0 | 0 | 0

8. Secondary Outcome: Incidence of Reoperation Due to Hematoma or Wound Dehiscence
Description: Number of subjects who underwent reoperation due to hematoma or wound dehiscence
Time Frame: Through day 60
Population: Safety analysis set: All subjects who received study drug treatment
Measure: Number; unit: participants
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 3 | 4 | 4
participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Incidence of Transfusion (Number of Units, Number of Units/Subject, Number of Subjects Transfused)
Time Frame: Day 60
Population: Efficacy analysis set: All subjects who received study drug and underwent planned surgery.
Measure: Number; unit: participants
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 3 | 4 | 4
participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With 90˚ Passive and Active Knee Flexion
Time Frame: 24, 48, and 72 hours
Population: Efficacy analysis set: All subjects who received study drug and underwent planned surgery.
Measure: Number; unit: participants
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 3 | 4 | 4
participants
  Number of subjects who had 90˚ active knee flexion at 24 hours | 0 | 0 | 0 | 0
  Number of subjects who had 90˚ active knee flexion at 48 hours | 0 | 0 | 0 | 1
  Number of subjects who had 90˚ active knee flexion at 72 hours | 1 | 0 | 0 | 0
  Number of subjects who had 90˚ passive knee flexion at 24 hours | 0 | 1 | 0 | 1
  Number of subjects who had 90˚ passive knee flexion at 48 hours | 1 | 0 | 0 | 1
  Number of subjects who had 90˚ passive knee flexion at 72 hours | 2 | 1 | 0 | 0

11. Secondary Outcome: Time to Complete Timed Up-and-Go (TUG) Test
Description: Physical therapy assessment (Timed Up-and-Go (TUG) test) was conducted once postsurgically on Day 1; at approximately 8:00 am and 8:00 pm (±2 hours) daily from Day 2 through hospital discharge; and on Day 7
Time Frame: Day 1; at approximately 8:00 am and 8:00 pm (±2 hours) daily from Day 2 through hospital discharge; and on Day 7
Population: Efficacy analysis set: All subjects who received study drug and underwent planned surgery.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 3 | 4 | 4
seconds
  Baseline | 16.4 (4.25) | 18.1 (10.73) | 14.6 (8.97) | 15.4 (6.92)
  Day 1: number analyzed (Participants) | 1 | 1 | 2 | 1
  Day 1 | 50.0 (NA) — 1 participant only | 80.0 (NA) — 1 participant only | 40.0 (7.07) | 80.0 (NA) — 1 participant only
  Day 2 - AM: number analyzed (Participants) | 2 | 2 | 3 | 1
  Day 2 - AM | 47.5 (10.61) | 90.0 (7.07) | 66.7 (23.63) | 85.0 (21.88)
  Day 2- PM: number analyzed (Participants) | 2 | 2 | 3 | 3
  Day 2- PM | 48.0 (14.14) | 85.0 (7.07) | 69.0 (25.94) | 41.0 (6.08)
  Day 2 -Discharge: number analyzed (Participants) | 3 | 3 | 4 | 2
  Day 2 -Discharge | 44.3 (6.03) | 51.1 (32.85) | 61.3 (31.76) | 40.0 (0.00)
  Day 7: number analyzed (Participants) | 4 | 3 | 3 | 1
  Day 7 | 28.4 (11.64) | 51.2 (32.89) | 32.3 (15.72) | 13.1 (NA) — 1 participant only

12. Secondary Outcome: Change in Knee and Thigh Measurements
Description: Leg difference in change from baseline is calculated by = (Operated Leg Change from Baseline) - (Non-Operated Leg Change from Baseline)
Time Frame: 48 hours and Day 7
Population: Efficacy analysis set: All subjects who received study drug and underwent planned surgery.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 3 | 4 | 4
cm
  Leg Difference in Change from Baseline in Thigh Circumference (cm) at 48 hours | 5.0 (4.73) | 6.7 (6.37) | 3.4 (4.54) | 6.1 (1.39)
  Leg Difference in Change from Baseline in Thigh Circumference (cm) at Day 7 | 4.3 (1.70) | 5.2 (6.17) | 0.8 (5.09) | 3.3 (3.18)
  Leg Difference in Change from Baseline in Knee Circumference at 48 hours | 4.1 (3.47) | 5.8 (5.37) | 2.2 (4.85) | 1.0 (5.25)
  Leg Difference in Change from Baseline in Knee Circumference at Day 7 | 2.6 (3.20) | 3.8 (8.25) | -1.4 (4.03) | 4.3 (0.35)

13. Secondary Outcome: Area Under the Curve (AUC) of NRS From 0-24 Hours, 0-48 Hours, and 24-48 Hours
Description: Numerical rating scale (NRS) at rest pain score (0 [no pain] to 10 [worst possible pain]) upon arrival at the PACU; at each in-hospital vital sign assessment beginning with the 2-hour assessment and ending with the 48-hour assessment; and the Day-7 follow-up visit. Summary is provided as area under the curve (AUC) of NRS from timepoint 0 to 24 hours, 0 to 48 hours, and 24 to 48 hours.
Time Frame: Preoperative; arrival in Post-Anesthesia Care Unit (PACU); 2, 4, 6, 8, 12, 16, 24, 36, 48 hours, Day 7
Population: Efficacy analysis set: All subjects who received study drug and underwent planned surgery.
Measure: Mean (Standard Deviation); unit: scores on a scale*hour
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
Number analyzed (Participants) | 4 | 3 | 4 | 4
scores on a scale*hour
  AUC(0-24) | 5230.0 (3416.48) | 4723.0 (3242.87) | 5119.3 (2587.32) | 6876.3 (2560.73)
  AUC(0-48) | 11375.1 (6159.89) | 12063.0 (3331.38) | 10859.5 (4761.97) | 13406.8 (5495.40)
  AUC(24-48) | 6145.1 (2786.30) | 7340.0 (1880.10) | 5740.3 (2244.90) | 6530.5 (2936.93)

ADVERSE EVENTS:
Time Frame: From screening to postsurgical day 60
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans whether or not considered drug-related. An AE could therefore have been any unfavorable and unintended sign (eg, abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug without any judgment about causality. Serious AEs were defined as per clinicaltrials.gov.
Arm/Group | DepoTXA 400mg | DepoTXA 800mg | DepoTXA 1200mg | IV Tranexamic Acid (TXA)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 2/3 | 4/4 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DepoTXA 400mg (N=4) | DepoTXA 800mg (N=3) | DepoTXA 1200mg (N=4) | IV Tranexamic Acid (TXA) (N=4)
Procedural pain (Injury, poisoning and procedural complications) | 3 | 2 | 3 | 2
Postprocedural hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Hypoesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was terminated on 27-Nov-2017 due to low enrollment; small sample sizes make data interpretation difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and investigator shall reasonably cooperate with Pacira to prepare abstract and manuscript reporting primary results within 90 and 120 days, respectively, of single and/or pooled analysis final CSR and shall publish no other trial results within 12 months after completion of final CSR. Institution shall submit all proposed written materials related to the trial ≥60 days before submission for presentation/publication. Pacira may embargo publication for an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT02922582/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT02922582/SAP_001.pdf